CLINICAL TRIAL: NCT06965114
Title: A Phase 1 Study of Combination Tovorafenib (DAY101) and Rituximab Treatment in Relapsed or Refractory Classical Hairy Cell Leukemia and Phase 2 Randomized Study Comparing Tovorafenib (DAY101) and Rituximab With Cladribine and Rituximab for Front-Line Treatment of Classical Hairy Cell Leukemia
Brief Title: Testing the Combination of Anti-cancer Drugs, Tovorafenib Plus Rituximab, in Patients With Hairy Cell Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-03281; NCI-2025-03281 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10664 (Other: Ohio State University Comprehensive Cancer Center LAO); 10664 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2025-05-08; First posted 2025-05-11 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Hairy Cell Leukemia; Recurrent Hairy Cell Leukemia; Refractory Hairy Cell Leukemia
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — Specimen Handling; Biopsy; Cladribine; Rituximab; CT-P10; tovorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1 (tovorafenib, rituximab) (Experimental): Patients receive tovorafenib PO QW for up to 16 weeks and rituximab IV QW on weeks 5-9 and 11, 13, and 15 in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, CT as clinically indicated, and bone marrow biopsy and aspiration throughout the study. Additionally, patients undergo buccal swab collection pre-study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Biological: Rituximab; Drug: Tovorafenib
- Phase 2 Arm A (cladribine, rituximab) (Active Comparator): Patients receive cladribine IV over 2 hours on days 1-5 of cycle 1 and rituximab IV on days 1, 8, 15, and 22 of cycles 2 and 3. Cycles repeat every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, CT as clinically indicated, and bone marrow biopsy and aspiration throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cladribine; Procedure: Computed Tomography; Biological: Rituximab
- Phase 2 Arm B (tovorafenib, rituximab) (Experimental): Patients receive tovorafenib PO on days 1, 8, 15, and 22 of each cycle and rituximab IV on days 1, 8, 15, and 22 of cycle 2 and on days 1 and 15 of cycles 3 and 4. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, CT as clinically indicated, and bone marrow biopsy and aspiration throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Biological: Rituximab; Drug: Tovorafenib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample and buccal swab collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
  Arms: Phase 2 Arm A (cladribine, rituximab)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Drug: Tovorafenib — Given PO
  Other Names: BIIB 024; BIIB-024; BIIB024; DAY 101; DAY-101; DAY101; MLN 2480; MLN-2480; MLN2480; Ojemda; pan-RAF Kinase Inhibitor DAY101; TAK 580; TAK-580; TAK580
  Arms: Phase 1 (tovorafenib, rituximab); Phase 2 Arm B (tovorafenib, rituximab)

SUMMARY:
This phase I/II trial tests the safety, side effects, and effectiveness of tovorafenib in combination with rituximab in patients with classical hairy cell leukemia (cHCL) that has come back after a period of improvement (recurrent) or that has not responded to previous treatment (refractory) and compares the effect of tovorafenib and rituximab to current standard treatment of cladribine and rituximab in cHCL patients that have not yet received treatment. Tovorafenib blocks certain proteins made by the mutated BRAF gene, which may help keep cancer cells from growing. It is a type of kinase inhibitor. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Cladribine damages the cell's deoxyribonucleic acid and may kill cancer cells. It is a type of antimetabolite. Giving tovorafenib in combination with rituximab may be safe and tolerable and more effective than cladribine with rituximab in treating patients with untreated, recurrent or refractory cHCL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of tovorafenib (DAY101) plus rituximab treatment in patients with relapsed or refractory classical hairy cell leukemia (cHCL). (Relapsed/Refractory Classical Hairy Cell Leukemia) II. To determine the minimal residual disease negative complete remission (MRD [-] CR) rate at completion of tovorafenib (DAY101) plus rituximab treatment versus cladribine plus rituximab for untreated cHCL. (Front-line Classical Hairy Cell Leukemia)

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. (Relapsed/Refractory Classical Hairy Cell Leukemia) II. To determine the overall response rate (ORR) and rate of minimal residual disease negative complete remission (MRD [-] CR) at completion of tovorafenib (DAY101) plus rituximab treatment for relapsed or refractory cHCL. (Relapsed/Refractory Classical Hairy Cell Leukemia) III. To determine the complete remission (CR) rate at completion of tovorafenib (DAY101) plus rituximab treatment in patients with relapsed or refractory cHCL. (Relapsed/Refractory Classical Hairy Cell Leukemia) IV. To estimate progression-free and overall survival after tovorafenib (DAY101) and rituximab treatment for patients with relapsed or refractory cHCL. (Relapsed/Refractory Classical Hairy Cell Leukemia) V. To determine the rate of durable CR after combination tovorafenib (DAY101) plus rituximab treatment, where durable CR is defined as achieving a CR and not experiencing relapse at 12 months after completing treatment. (Front-line Classical Hairy Cell Leukemia) VI. To determine the safety of the combination of tovorafenib (DAY101) plus rituximab. (Front-line Classical Hairy Cell Leukemia) VII. To determine the clonal evolution of cHCL at the time of relapse by whole exome sequencing (WES) and ribonucleic acid sequencing (RNAseq). (Front-line Classical Hairy Cell Leukemia)

EXPLORATORY OBJECTIVES:

I. To evaluate mitogen-activated protein kinase (MAPK) activation status pre- and post-treatment in peripheral blood circulating cells (multiple timepoints during cycle 1: pre-dose [cycle (C) 1 day (D) 1], at 24 [C1D2] and 72 [C1D4] hours after first dose of tovorafenib [DAY101] and pre-dose on C1D8) to demonstrate that the drug did what it is expected to do and to assess the kinetics of phosphorylated-extracellular signal-regulated kinase (pERK) clearance. (Front-line Classical Hairy Cell Leukemia) II. To describe changes in T- and natural killer (NK)-cell function prior to, after tovorafenib (DAY101) single agent treatment, and after tovorafenib (DAY101) plus rituximab combination treatment in patients with cHCL. (Front-line Classical Hairy Cell Leukemia) III. To identify mutations or changes in transcription profile through whole exome and RNA sequencing of leukemia cell samples at baseline and at time of relapse after combination treatment, which can be used to guide analysis in larger cohorts or with future functional studies to determine mechanisms of resistance (or sensitivity) to the therapy. (Front-line Classical Hairy Cell Leukemia)

OUTLINE:

PHASE 1: Patients receive tovorafenib orally (PO) once weekly (QW) for up to 16 weeks and rituximab intravenously (IV) QW on weeks 5-9 and 11, 13, and 15 in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, computed tomography (CT) as clinically indicated, and bone marrow biopsy and aspiration throughout the study. Additionally, patients undergo buccal swab collection pre-study.

PHASE 2: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive cladribine IV over 2 hours on days 1-5 of cycle 1 and rituximab IV on days 1, 8, 15, and 22 of cycles 2 and 3. Cycles repeat every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, CT as clinically indicated, and bone marrow biopsy and aspiration throughout the study.

ARM B: Patients receive tovorafenib PO on days 1, 8, 15, and 22 of each cycle and rituximab IV on days 1, 8, 15, and 22 of cycle 2 and on days 1 and 15 of cycles 3 and 4. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, CT as clinically indicated, and bone marrow biopsy and aspiration throughout the study.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of classical hairy cell leukemia (HCL), including demonstration of BRAF V600E mutation by immunohistochemistry, molecular diagnostic testing, or polymerase chain reaction (PCR)
* PHASE 1 ONLY: Prior therapy with at least one purine nucleoside analog-containing regimen (fludarabine, pentostatin, or cladribine) unless contraindicated. Prior vemurafenib alone is allowed in the relapsed/refractory cohort
* PHASE 2 ONLY: No prior HCL-directed treatment for front-line cohort. The design of this cohort is such that the patients will need to be treatment naïve
* Age ≥ 18 years. Because no dosing or adverse event (AE) data are currently available on the use of tovorafenib (DAY101) or cladribine in combination with rituximab in patients < 18 years of age, children are excluded from this study
* Patients must meet indications for treatment of cHCL:

  * Absolute neutrophil count < 1,000/mcL
  * Platelets < 100,000/mcL
  * Hemoglobin < 10 g/dL
  * Recurrent infections
  * Symptomatic and/or progressive extramedullary disease including lymph nodes and bone lesions
  * Progressive or symptomatic splenomegaly or hepatomegaly
  * Disease-related constitutional symptoms consisting of unexplained weight loss exceeding 10% body weight during the preceding 6 months, Cancer Therapy Evaluation Program (CTEP) active version of the Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or 3 fatigue, and/or fever > 100.5 F or night sweats for > 2 weeks without evidence of active infection
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%); ECOG performance status > 2 (Karnofsky < 60%) will be allowed if considered due to HCL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN (unless related to Gilbert's disease or HCL; patients with documented Gilbert's disease may be enrolled with sponsor approval provided total bilirubin is ≤ 2.0 x ULN)
* Creatinine clearance (ClCr) ≥ 30 mL/min
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load for > 6 months
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Electrocardiogram (ECG) without evidence of clinically significant ventricular arrhythmias or ischemia as determined by the investigator and a rate-corrected QT interval (QTc, Bazett's formula) of < 480 msec
* The effects of tovorafenib (DAY101), cladribine, and rituximab on the developing human fetus are unknown. For this reason and because BRAF kinase inhibitor agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential (WOCBP) and men must agree to use two forms of adequate contraception (including a highly effective birth control method in addition to a barrier method) during treatment prior to study entry and for the duration of study treatment participation and 12 months after the last dose of the study medication

  * WOCBP should use effective non-hormonal contraception during treatment and for 12 months after the last dose of the study medication. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. For male patients with a female partner of childbearing potential, a condom should be used for contraception in addition to one of the highly effective contraception methods prior to the study, for the duration of study treatment, and 12 months after the last dose of the study medication. Male patients must not father a child or donate sperm while participating in this study
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives (LARs) may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Central nervous system (CNS) involvement with HCL is very rare, and therefore the biology of the disease in patients with CNS involvement may not be representative of the disease under study as a whole. Patients with treated brain metastases are eligible if follow-up brain imaging after CNS-directed therapy shows no evidence of progression
* Patients with HCL who are BRAF V600E mutation negative and those with the variant HCL
* Patients with platelets < 50,000/mCL
* Patients on warfarin and direct oral anticoagulants (due to risk of bleeding)
* Patients who have not recovered from AEs as a result of prior anti-cancer therapy (i.e., have residual toxicities > grade 1), with the exception of alopecia
* Patients who are receiving any other investigational agents
* Patients who are receiving strong CYP2C8 inhibitors, inducers, and breast cancer resistance protein (BCRP) substrates with narrow therapeutic index
* Patients who are pregnant, breastfeeding, and/or unwilling to use adequate contraception during the study period and for 12 months after completion of the study
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to tovorafenib (DAY101) or other agents used in the study, including those with a previous history of severe infusion-related reaction (anaphylaxis) with rituximab administration
* Patients with known hypersensitivity to any of the study drugs
* Patients with an inability to swallow oral medications or with gastrointestinal impairment
* Live or live-attenuated vaccines within 28 days of randomization
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because tovorafenib (DAY101) is a BRAF kinase inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with tovorafenib (DAY101), breastfeeding should be discontinued if the mother is treated with tovorafenib (DAY101). These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-06-27 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (Phase 1) | During cycles 1-3 (cycle length = 28 days)
  Adverse events (AEs) will be documented and summarized by type, grade, severity, and attribution using the Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 criteria for non-hematologic toxicities and table of criteria for hematologic toxicities. In addition, the number of treatment cycles received and reasons for going off treatment will be summarized to assess treatment tolerability. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Minimal residual disease negative complete remission (MRD [-] CR) rate (Phase 2) | At completion of tovorafenib plus rituximab treatment versus cladribine plus rituximab
  Will be calculated as the proportion of patients who achieve MRD (-) CR to therapy divided by the total number of patients for each treatment arm. All randomized patients or evaluable patients will be included in calculating the rate of MRD (-) CR for the study along with corresponding 95% binomial confidence intervals (CIs) (assuming that the number of patients who respond is binomially distributed). The MRD (-) CR rate will be compared between the untreated classical hairy cell leukemia (cHCL) patients with tovorafenib plus rituximab treatment and the patients with cladribine plus rituximab using the chi-square test or Fisher's exact test.

SECONDARY OUTCOMES:
MRD (-) CR rate (Phase 1) | At completion of tovorafenib plus rituximab
  Will be calculated along with corresponding 95% binomial CIs (assuming that the number of patients who respond is binomially distributed).
Overall response rate (ORR) (Phase 1) | At completion of tovorafenib plus rituximab
  Will be calculated along with corresponding 95% binomial CIs (assuming that the number of patients who respond is binomially distributed). For the phase 2 portion, the ORR will be compared between the untreated cHCL patients with tovorafenib plus rituximab treatment and the patients with cladribine plus rituximab using the chi-square test or Fisher's exact test.
Progression-free survival (Phase 1) | From initiation of therapy to documented progression or death without progression, assessed up to 10 years
  Will initially be modeled using Kaplan-Meier methods, resulting in median survival times with 95% CI, assuming sufficient events have occurred.
Overall survival (Phase 1) | From initiation of therapy to death from any cause, assessed up to 10 years
  Will initially be modeled using Kaplan-Meier methods, resulting in median survival times with 95% CI, assuming sufficient events have occurred.
Incidence of AEs (Phase 2) | From first dose of study treatment up to 30 days after the last dose of study medication, or until the start of subsequent antineoplastic therapy, whichever occurs first
  Will be documented and summarized by type, grade, severity, and attribution using the CTCAE v 5.0 criteria for non-hematologic toxicities and the table on Criteria for Hematologic Toxicities. Will review all AE data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The incidence of severe (grade 3+) AEs or toxicities will be described. The number of treatment cycles received and reasons for going off treatment will be summarized to assess treatment tolerability. Will assess tolerability of the regimens through assessing the number of patients who required dose modifications and/or dose delays. Tolerability measures will be assessed within each treatment arm, and will explore differences in these measures between the arms. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Rate of durable complete remission (CR) (Phase 2) | Up to 12 months after completing treatment
  Will be defined as achieving a CR and not experiencing relapse at 12 months after completing treatment.
Mutations or changes in transcription profile (Phase 1) | At baseline and at time of relapse, assessed up to 10 years
  Will be assessed using whole exome and ribonucleic acid sequencing.

OTHER OUTCOMES:
Mitogen-activated protein kinase activation status (Phase 1) | During cycle 1 (cycle length = 28 days)
  Graphical analyses will be largely used to assess potential patterns and relationships. All continuous measurements will be summarized using mean with standard deviations or median with range at each time point. Changes in these measurements from baseline to after treatment or baseline to progression will be assessed using paired t-tests or corresponding bob-parametric tests. The changes will also be compared between the treatment groups using two sample t-tests or Wilcoxon tests.
Changes in T and natural killer cell function (Phase 1) | Prior to and after tovorafenib and after tovorafenib plus rituximab, assessed up to 10 years
  Graphical analyses will be largely used to assess potential patterns and relationships. All continuous measurements will be summarized using mean with standard deviations or median with range at each time point. Changes in these measurements from baseline to after treatment or baseline to progression will be assessed using paired t-tests or corresponding bob-parametric tests. The changes will also be compared between the treatment groups using two sample t-tests or Wilcoxon tests.

CONTACTS AND LOCATIONS:
Overall Officials: Seema A Bhat, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO
Locations (1):
- Ohio State University Comprehensive Cancer Center LAO, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm